CLINICAL TRIAL: NCT05662410
Title: Choroidal Morphology Changes After Aflibercept Therapy in Pachychoroid Neovasculopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kim's Eye Hospital (Other)
Collaborators: Nune Eye Hospital, Seoul, Korea (Other); HanGil Eye Hospital (Other)
Responsible Party: Principal Investigator, Jae Hui Kim, Principle Investigator, Kim's Eye Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-10-001
Record Dates: First submitted 2022-12-07; First posted 2022-12-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Pachychoroid Neovasculopathy
Keywords: Pachychoroid neovasculopathy; Aflibercept; Choroidal morphology

STUDY DESIGN:
Intervention Model Description: Three monthly injections of intravitreal aflibercept during the first 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aflibercept treatment group (Experimental): Patients receiving three monthly aflibercept injections
  Interventions: Drug: Three monthly injections of intravitreal aflibercept

INTERVENTIONS:
Drug: Three monthly injections of intravitreal aflibercept — Three monthly intravitreal injection of aflibercept (2.0mg / 0.05ml) after diagnosis of pathychoroid neovasculopathy.

SUMMARY:
In the present study, investigators attempt to evaluate the short-term, detailed changes in choroidal morphology after three monthly injections of aflibercept in pachychoroid neovasculopathy. The association between these changes and clinical outcomes will be additionally investigated. The primary purpose of this study is to provide reference data regarding the aflibercept-related morphologic changes that implicate structural and functional choroidal alteration, and hence its clinical implications.

DETAILED DESCRIPTION:
Pachychoroid neovasculopathy (PNV), is a recently proposed entity after advancements in retinal imaging, belonging to the pachychoroid spectrum of diseases. It is a prevalent subtype of neovascular age-related macular degeneration (AMD) in the Asian population (19.5%~41.6% among neovascular AMD), characterized by presence of type 1 macular neovascularization (MNV) without polypoidal lesion in an eye exhibiting pachychoroid features, although its pathogenesis is not fully understood. In addition, PNV can be distinguished from typical neovascular AMD by a relative absence of drusen or pseudodrusen, younger age of onset, and thickened choroid with pachyvessels. Although both neovascular AMD and PNV respond well to anti-vascular endothelial growth factor (VEGF) therapy, separate analysis of treatment outcomes in PNV merits further investigation targeting the different underlying pathologies.

It is well-known that anti-VEGF therapy influences choroidal structures, including choroidal thickness, choroidal vascularity index, and choroidal area. In general, decrease in choroidal thickness after aflibercept injection is more prominent than that after ranibizumab or bevacizumab injections. Some investigators postulated that this difference in the effect on choroid is responsible for the superior efficacy of aflibercept in polypoidal choroidal vasculopathy (PCV) over other anti-VEGF agents and influence the choice of anti-VEGF agent in real-world practice. To date, several investigators have demonstrated changes in choroidal thickness after anti-VEGF therapy in PNV. However, the detailed changes in choroidal morphology after aflibercept therapy and its clinical implications in pachychoroidal neovasculopathy remain to be elucidated.

In the present study, investigators attempt to evaluate the short-term, detailed changes in choroidal morphology after three monthly injections of aflibercept in pachychoroid neovasculopathy. The association between these changes and clinical outcomes will be additionally investigated. The primary purpose of this study is to provide reference data regarding the aflibercept-related morphologic changes that implicate structural and functional choroidal alteration, and hence its clinical implications.

ELIGIBILITY:
Inclusion Criteria:

* Willing, committed, and able to return for all clinic visits and complete all study related procedures.
* Able to read, (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or a family member) understand and willing to sign the informed consent form.
* Signed informed consent
* Patients aged 50 years or older
* Patients diagnosed with treatment naïve pachychoroid neovasculopathy

  * Diagnostic criteria of PNV

    1. Presence of type 1 MNV
    2. Subfoveal choroidal thickness ≥250 µm
    3. Focal or diffuse choroidal thickening
    4. Presence of dilated choroidal vessels (pachyvessels)
    5. Thinning or absence of choriorapillaris and Sattler's layer overlying pachyvessels
    6. Absence of drusen or pseudodrusen, except for pachydrusen
* ETDRS BCVA letter score ≥25 letters (approximately 20/320 or better) in the study eye

Exclusion Criteria:

* Any prior ocular (in the study eye) or systemic treatment or surgery for neovascular AMD except dietary supplements or vitamins.
* Prior treatment with anti-VEGF agents
* Known serious allergy to the fluorescein sodium for injection in angiography.
* Significant media opacities, including cataract, in the study eye that might interfere with visual acuity, assessment of safety, or fundus photography.
* Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the patient beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.
* Any ocular or periocular infection within the last 2 weeks prior to Screening in either eye.
* Any history of uveitis in either eye.
* Presence of definite chorioretional anastomosis
* Subretinal hemorrhage that is either 50% or more of the total lesion area, or if the blood is under the fovea and is 1 or more disc areas in size in the study eye. (If the blood is under the fovea, then the fovea must be surrounded 270 degrees by visible choroidal neovascularization.)
* Scar or fibrosis, making up > 50% of total lesion in the study eye.
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Presence of retinal pigment epithelial tears or rips involving the macula in the study eye.
* History or clinical evidence of diabetic retinopathy, diabetic macular edema or any other vascular disease affecting the retina, other than AMD, in either eye.
* Any concurrent intraocular condition in the study eye (e.g. cataract) that, in the opinion of the investigator, could require either medical or surgical intervention during the 76 week study period.
* Prior vitrectomy in the study eye
* Any history of macular hole of stage 2 and above in the study eye.
* Any intraocular or periocular surgery within 3 months of Day 1 on the study eye, except lid surgery, which may not have taken place within 1 month of day 1, as long as its unlikely to interfere with the injection.
* Prior trabeculectomy or other filtration surgery in the study eye.
* Uncontrolled glaucoma (defined as intraocular pressure ≥ 25 mmHg despite treatment with antiglaucoma medication) in the study eye.
* Active intraocular inflammation in either eye.
* Active ocular or periocular infection in either eye.
* Aphakia or pseudophakia with absence of posterior capsule (unless it occurred as a result of a yttrium aluminum garnet posterior capsulotomy) in the study eye.
* History of corneal transplant or corneal dystrophy in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-26 (Actual)

PRIMARY OUTCOMES:
Area of choroidal layer | Baseline and Week 12
  Change in the area of each choroidal layer from baseline to week 12. The area will be assessed based on optical coherence tomography (OCT) image.

SECONDARY OUTCOMES:
Subfoveal choroidal thickness | Baseline and Week 12
  Changes in subfoveal choroidal thickness from baseline to week 12. The thickness will be assessed based on OCT image
Largest choroidal vessel diameter | Baseline and Week 12
  Changes in the largest choroidal vessel diameter from baseline to week 12. The diameter will be assessed based on OCT image
Choroidal vascularity index (CVI) | Baseline and Week 12
  Changes in choroidal vascularity index from baseline to week 12. The CVI will be assessed based on OCT image
Lesion size | Baseline and Week 12
  Changes in lesion size on OCT-angiography from baseline to week 12. The lesion size will be assessed based on OCT angiography image
Best-corrected visual acuity (BCVA) | Baseline and Week 12
  Changes in BCVA from baseline to week 12. The BCVA will be assessed using manifest refraction with early treatment of diabetic retinopathy score chart
Fluid after loading injections | Baseline and Week 12
  Resolution of fluid after loading injections from baseline to week 12. The resolution will be assessed based on OCT image
Choroidal morphology changes | Baseline and Week 12
  Difference in choroidal morphology changes between patients with and without fluid resolution. The morphology changes will be assessed based on OCT image
Central retinal thickness | Baseline and Week 12
  Changes in central retinal thickness (CRT) from baseline to week 12. The CRT will be assessed based on OCT image.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hui H Kim, M.D., Principal Investigator — Kim's Eye Hospital, South Korea
Locations (1):
- Jae Hui Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pang CE, Freund KB. Pachychoroid neovasculopathy. Retina. 2015 Jan;35(1):1-9. doi: 10.1097/IAE.0000000000000331. PMID 25158945
- [Background] Cheung CMG, Lee WK, Koizumi H, Dansingani K, Lai TYY, Freund KB. Pachychoroid disease. Eye (Lond). 2019 Jan;33(1):14-33. doi: 10.1038/s41433-018-0158-4. Epub 2018 Jul 11. PMID 29995841
- [Background] Pellegrini M, Bernabei F, Mercanti A, Sebastiani S, Peiretti E, Iovino C, Casini G, Loiudice P, Scorcia V, Giannaccare G. Short-term choroidal vascular changes after aflibercept therapy for neovascular age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 2021 Apr;259(4):911-918. doi: 10.1007/s00417-020-04957-5. Epub 2020 Oct 13. PMID 33048236
- [Background] Kim JH, Lee TG, Chang YS, Kim CG, Cho SW. Short-term choroidal thickness changes in patients treated with either ranibizumab or aflibercept: a comparative study. Br J Ophthalmol. 2016 Dec;100(12):1634-1639. doi: 10.1136/bjophthalmol-2015-308074. Epub 2016 Mar 7. PMID 26951770
- [Background] Padron-Perez N, Arias L, Rubio M, Lorenzo D, Garcia-Bru P, Catala-Mora J, Caminal JM. Changes in Choroidal Thickness After Intravitreal Injection of Anti-Vascular Endothelial Growth Factor in Pachychoroid Neovasculopathy. Invest Ophthalmol Vis Sci. 2018 Feb 1;59(2):1119-1124. doi: 10.1167/iovs.17-22144. PMID 29490349
- [Background] Schworm B, Luft N, Keidel LF, Kreutzer TC, Herold TR, Priglinger SG, Siedlecki J. Vanishing pachy-choroid in pachychoroid neovasculopathy under long-term anti-vascular endothelial growth factor therapy. BMC Ophthalmol. 2021 Jun 30;21(1):269. doi: 10.1186/s12886-021-02022-1. PMID 34193089
- [Background] Jung BJ, Kim JY, Lee JH, Baek J, Lee K, Lee WK. Intravitreal aflibercept and ranibizumab for pachychoroid neovasculopathy. Sci Rep. 2019 Feb 14;9(1):2055. doi: 10.1038/s41598-019-38504-y. PMID 30765771